CLINICAL TRIAL: NCT06544239
Title: Virtual Reality Basketball Asymmetric Training
Brief Title: Virtual Reality Asymmetric Training of Technology And Tactics for Professional Basketball Players
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Man Yuan, Researcher, Student of Faculty Education, Dr., Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: University Putra Malaysia FPP
Record Dates: First submitted 2024-07-06; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Asymmetric Limb Muscle Stiffness; Recovery, Psychological; Body Schema
Keywords: Virtual Reality Training; Physical; Recovery; Sports Psychology; Skill

STUDY DESIGN:
Intervention Model Description: Experimental Group (virtual reality training) & Control Group (traditional training)
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual reality basketball asymmetric training (Experimental)
  Interventions: Behavioral: Virtual reality basketball asymmetric training
- Traditional basketball asymmetric training (Experimental)
  Interventions: Behavioral: Traditional basketball asymmetric training

INTERVENTIONS:
Behavioral: Virtual reality basketball asymmetric training — This study established two experimental groups, namely the experimental group and the control group. The experimental group received virtual reality device assisted training, while the control group received traditional training
  Arms: Virtual reality basketball asymmetric training
Behavioral: Traditional basketball asymmetric training — This study established two experimental groups, namely the experimental group and the control group. The experimental group received virtual reality device assisted training, while the control group received traditional training
  Arms: Traditional basketball asymmetric training

SUMMARY:
This study exploring the effects of virtual reality basketball asymmetric training on the technical and tactical ability of professional basketball players (male and female) through the use of virtual reality devices.

DETAILED DESCRIPTION:
The experimental conclusion of this study was obtained by comparing virtual reality basketball asymmetric training with traditional basketball asymmetric training (using cRCT random experimental grouping)

ELIGIBILITY:
Inclusion Criteria:

* Asymmetric limbs
* Psychological defects
* Joint stiffness
* Amyotrophic lateral sclerosis

Exclusion Criteria:

* Physically and mentally healthy individuals
* Schizophrenia patients
* Cognitive impairment patients

Ages: 17 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-10 (Estimated)

PRIMARY OUTCOMES:
Effects of Asymmetric Training in Virtual Reality Basketball on The Complex Technical Completion Scores of Professional Basketball players | Pretest：July 27th Post-test 1：August 25th Post-test 2：September 22nd
  Examine the effect of virtual reality training across pretest, post-test 1, and post-test 2 on asymmetrical scores of complex technical abilities in terms of professional basketball players' dribbling, driving, passing, and rebounding in China.
  This study used DJ Osmo Action 3 camera and GoPose software to capture, measure, and analyze the basketball technique movements of the experimental subjects. The specific measurements are listed below： Technical Completion Rate (0/100 points) Technical Connection Rate (0/100 points)
Effects of Asymmetric Training in Virtual Reality Basketball on The Complex Technical Completion Rate of Professional Basketball players | Pretest：July 27th Post-test 1：August 25th Post-test 2：September 22nd
  Examine the effect of virtual reality training across pretest, post-test 1, and post-test 2 on asymmetrical rate of complex technical abilities in terms of professional basketball players' shooting, layup and defensive in China.
  This study used DJ Osmo Action 3 camera and GoPose software to capture, measure, and analyze the basketball technique movements of the experimental subjects. The specific measurements are listed below： Technical Accuracy Rate (%) Technology Success Rate (%)
Effects of Asymmetric Training in Virtual Reality Basketball on Complex Tactics Scores of Professional Basketball Players | Pretest：July 27th Post-test 1：August 25th Post-test 2：September 22nd
  Examine the effect of virtual reality training across pretest, post-test 1, and post-test 2 on asymmetrical scores level of tactical abilities in terms of professional basketball players' 3-man organized offense, 3-man organized defense, 4-man organized offense, 4-man organized defense, 5-man organized offense and 5-man organized defense in China.
  This study used DJ Osmo Action 3 camera and Dartfish software to capture, measure, and analyze the basketball tactical execution process of the experimental subjects. The specific measurements are listed below： Tactical Completion Rate (0/100 points) Tactical Connection (0/100 points) Tactical Decision-making Ability (0/100 points) Tactical Selection Accuracy (0/100 points) Tactical SuccessRate (0/100 points)

CONTACTS AND LOCATIONS:
Overall Officials: Soh Kim Geok, Professor, Study Chair — Universiti Putra Malaysia Research Institute Branch
Locations (1):
- Shandong Provincial Sports Training Center, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided